CLINICAL TRIAL: NCT01647763
Title: Hemorrhoidal Artery Ligation and Rectoanal Repair Versus Stapled Hemorrhoidopexy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Lukas Marti, Leitender Arzt (attending surgeon), Cantonal Hospital of St. Gallen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EKSG11/042
Record Dates: First submitted 2012-07-18; First posted 2012-07-24 (Estimated); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Hemorrhoids
Keywords: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids | interventions — Retinoic Acid Receptor alpha

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- HAL/RAR (Experimental): hemorrhoidal artery ligation with rectoanal repair
  Interventions: Procedure: Hemorrhoidal artery ligation with rectoanal repair
- Stapled hemorrhoidopexy (Active Comparator): procedure for prolapse and hemorrhoids (PPH)
  Resection using a circular stapler
  Interventions: Procedure: Stapled hemorrhoidopexy

INTERVENTIONS:
Procedure: Hemorrhoidal artery ligation with rectoanal repair — Hemorrhoidal arteries will be detected using an ultrasound Doppler probe. The arteries will be sutured with at least 4 Z-sutures.
  In the area with the 3 largest knots a purse string suture will be placed.
  Other Names: HAL (hemorrhoidal artery ligation); RAR (rectoanal repair)
  Arms: HAL/RAR
Procedure: Stapled hemorrhoidopexy — A purse string suture will be placed just below the hemorrhoidal cushion. Fixing the suture around the shaft of a circular PPH 03 stapler (Ethicon Endo-Surgery). Hemorrhoids will be removed by firing the stapler. Sufficiency of the stapler line will be examined through a proctoscope. Eventual sources of bleeding will be sutured.
  Other Names: Longo procedure
  Arms: Stapled hemorrhoidopexy

SUMMARY:
Background:

Hemorrhoids of grade 3 and 4 can be treated either by conventional, rather invasive procedures, like Milligan-Morgan or Ferguson or by modern, less invasive procedures with less postoperative pain. Doppler guided hemorrhoidal artery ligation and stapled hemorrhoidopexy are examples for such modern procedures. Hemorrhoidal artery ligation causes less post operative pain than stapled hemorrhoidopexy, however the former has a higher recurrence rate. Combining hemorrhoidal artery ligation with rectoanal repair should reduce the recurrence rate without increasing the post operative pain.

Hypothesis and aim:

The study tries to prove the assumption that combined hemorrhoidal artery ligation and rectoanal repair cause less pain and have less post operative complications than stapled hemorrhoidopexy.

ELIGIBILITY:
Inclusion Criteria:

* hemorrhoids grade 3
* no active anti-coagulation treatment
* no hemorrhoidal recurrence
* no previous surgery on rectum or anus
* no previous local radiotherapy
* no mental incapacities, good study compliance can be expected
* no severe incontinence (Wexner score > 12)
* no severe comorbidities
* no inflammatory anal diseases (abscesses, fistulas)
* informed consent

Exclusion Criteria:

* patient wish
* inoperability with the assigned intervention, switching to other treatment method

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2011-07 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Pain POD1 | between 6:00 am and 8:00 am the day after surgery
  Visual analogue scale (VAS).
  Additionally recording of the pain medication used.

SECONDARY OUTCOMES:
Pain after 8h | 8 hours after surgery
  Measuring post operative pain using the visual analogue scale (0 - 10).
  Additionally recording of the pain medication used.
Pain 30d | 30 days after surgery
  visual analogue scale
Pain 1y | 1 year after surgery
  visual analogue scale
Pain 2y | 2 years after surgery
  visual analogue scale
post operative surgical complications | within 30 post operative days
  Number and severity according to the Dindo classification (Ann Surg 240:205)
duration of medical leave | up to 3 months after surgery
  data will be obtained from primary care physician
Continence 30d | 30 days after surgery
  Physician obtains data to calculate the Wexner Score (Dis Colon Rectum 36:77).
  Score will be compared with pre-operative score.
Continence 1y | 1 year after surgery
  Wexner score
Continence 2y | 2 years after surgery
  Wexner score
  Additionally anorectal manometry (results will be compared with pre-operative data).

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Marti, MD, Principal Investigator — Cantonal Hospital St. Gallen, Department of Surgery
Locations (2):
- Switzerland (2):
  - Kantonsspital Rorschach, _Rorschach
  - Kantonsspital St. Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of the Department of Surgery (in German only) — http://www.chirurgie.kssg.ch/home/unsere_klinik/Leistungsangebot_standort_st_gallen/koloproktologie.html